CLINICAL TRIAL: NCT00593957
Title: Trial of Dextromethorphan in Rett Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study changed to a placebo controlled trial of dextromethorphan
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, SakkuBai Naidu, M.D., Professor of Neurology and Pediatrics, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FD2408
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2013-07

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Dextromethorphan
MeSH Terms: conditions — Rett Syndrome | interventions — Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DM1( 0.25 mg/kg /day) (Experimental): Dextromethorphan 0.25 mg/kg per day
  Interventions: Drug: Dextromethorphan
- DM2 (2.5 mg/kg/day) (Experimental): Dextromethorphan 2.5 mg/kg/day
  Interventions: Drug: Dextromethorphan
- DM3 (5mg/kg/day) (Experimental): Dextromethorphan 5mg/kg/day
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — Subjects will be randomized to receive one of three dosage groups either 0.25 mg/kg per day; or 2.5 mg/kg/day; or 5mg/kg/day of Dextromethorphan Polistirex (Delsym)oral syrup, which will be given exactly 12 hours apart in two divided doses during the 6 month trial.
  Other Names: Delsym
Drug: Dextromethorphan — Dextromethorphan polistirex. Doses are 0.25 mg/kg/day, 2.5mg/kg/day, and 5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months.
  Other Names: Delsym

SUMMARY:
Increased brain glutamate and its N-methyl-D-aspartate (NMDA) receptors found in the brain of younger Rett syndrome (RTT) patients cause toxic damage to neurons (the brain's nerve cells), and contributing to EEG spikes. Dextromethorphan (DM) acts by blocking NMDA/glutamate receptors. This study is being done to determine if DM will prevent the harmful over-stimulation of the neurons thereby reducing EEG spike activity. Treatment with DM consists of one of 3 different doses (0.25 mg/kg per day; or 2.5 mg/kg/day; or 5mg/kg/day), and aims to find out which dose if any will help improve EEG abnormalities, behavior, cognition, and reduce seizures, as well as improve breathing abnormalities, motor capabilities, bone density, and GI dysfunction.

The study will include 90 females and males with RTT, 2 years-14.99 years of age, with a mutation in the methyl CpG binding protein 2 (MECP2) gene, and spikes on EEG, with or without clinical seizures.

DETAILED DESCRIPTION:
Patients meeting eligibility criteria(mutation +ve and having EEG spikes), will be admitted to the Pediatric Clinical Research Unit at Johns Hopkins Hospital and will have pharmacokinetics of DM determined to establish that they are rapid metabolizers of the drug. The baseline studies on initial admission include neurological, neuropsychology,EEG, gastroenterology, Occupational and Physical therapy evaluations. If the subject is a rapid metabolizer they will be randomized to one of the three drug doses. They are contacted by telephone, weekly in the first month, and monthly thereafter. They will be examined by a neurologist at 2 weeks,1 month, and 3 months during the drug trial. At each of these visits they will also be monitored for changes in complete blood count (CBC), electrolytes, and EKG. At the end of the 6 month drug trial the patients will be readmitted to Johns Hopkins Hospital when all baseline studies are repeated. Cost of travel, hospitalization and interim tests are free to participants.

ELIGIBILITY:
Inclusion Criteria:

1. those who have classic or atypical RTT with a proven mutation in the MeCP2 gene;
2. those with documented EEG evidence of spike activity who may or may not have clinical seizures;
3. subjects must be between 2years -14.99 years of age.

Exclusion Criteria:

1. those without an established mutation in the MeCP2 gene;
2. those who do not have EEG evidence of spike activity;
3. those with mutations in the MeCP2 gene but who have had brain resection or surgical intervention; for example, tumor, hydrocephalus, severe head trauma; or, an associated severe medical illnesses such as vasculopathies, malignancies, diabetes, thyroid dysfunction, etc;
4. those on medications that could interact with DM, e.g. monoamine oxidase (MAO) inhibitors, selective serotonin reuptake inhibitor (SSRI), sibutramine etc. to avoid a serotonin syndrome; quinidine and drugs metabolized by the Cytochrome P450 (CYP450) isoform cytochrome P450 2D6 (CYP2D6) (e.g. amiodarone, haloperidol, propafenone, thioridazine);
5. those proven to be intermediate or slow metabolizers of DM;
6. those with reported adverse reactions to DM;
7. those whose pregnancy test is positive; and,
8. those showing poor compliance with any aspect of the study;
9. foster children

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2004-08; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SakkuBai Naidu, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute/Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 2004 to 2010. Study initiation was delayed due to the closure of Johns Hopkins Medicine Institutional Review Board(JHMIRB). Patients were recruited from our Kennedy Krieger Institute (KKI)medical clinics, physician referrals,and parent organizations. Parents were sent letters of invitation.
Pre-assignment Details: Pharmacokinetics in enrolled subjects required her to be a fast metabolizer of Dextromethorphan (DM).
Groups:
- DM1( 0.25 mg/kg /Day): Dextromethorphan 0.25 mg/kg per day
  Dextromethorphan : Dextromethorphan polistirex. Doses are 0.25 mg/kg/day, 2.5mg/kg/day, and 5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months.
  Dextromethorphan : Subjects will be randomized to receive one of three dosage groups either 0.25 mg/kg per day; or 2.5 mg/kg/day; or 5mg/kg/day of Dextromethorphan Polistirex (Delsym)oral syrup, which will be given exactly 12 hours apart in two divided doses during the 6 month trial.
- DM2 (2.5 mg/kg/Day): Dextromethorphan 2.5 mg/kg/day
  Dextromethorphan : Dextromethorphan polistirex. Doses are 0.25 mg/kg/day, 2.5mg/kg/day, and 5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months.
  Dextromethorphan : Subjects will be randomized to receive one of three dosage groups either 0.25 mg/kg per day; or 2.5 mg/kg/day; or 5mg/kg/day of Dextromethorphan Polistirex (Delsym)oral syrup, which will be given exactly 12 hours apart in two divided doses during the 6 month trial.
- DM3 (5mg/kg/Day): Dextromethorphan 5mg/kg/day
  Dextromethorphan : Dextromethorphan polistirex. Doses are 0.25 mg/kg/day, 2.5mg/kg/day, and 5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months.
  Dextromethorphan : Subjects will be randomized to receive one of three dosage groups either 0.25 mg/kg per day; or 2.5 mg/kg/day; or 5mg/kg/day of Dextromethorphan Polistirex (Delsym)oral syrup, which will be given exactly 12 hours apart in two divided doses during the 6 month trial.
Period: Overall Study
Arm/Group | DM1( 0.25 mg/kg /Day) | DM2 (2.5 mg/kg/Day) | DM3 (5mg/kg/Day)
Started | 13 | 13 | 12
Completed | 13 | 12 | 10
Not Completed | 0 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DM1( 0.25 mg/kg /Day) | DM2 (2.5 mg/kg/Day) | DM3 (5mg/kg/Day) | Total
Number analyzed (Participants) | 13 | 13 | 12 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 12 | 38
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.54 (2.70) | 6.31 (3.50) | 6.08 (3.06) | 6.32 (3.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 12 | 38
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Difference in EEG Spike Counts at Six Months Compared to Baseline for Each Treatment Arm.
Description: Difference in EEG spike count means pre and 6 months post-treatment in each of three treatment groups.
Time Frame: Initial and 6-month post-treatment
Population: 33/35 participants who completed the protocol with two epochs of 5 mins of non-Rapid eye movement (REM)sleep during which spikes could be counted pre and post DM intake.
Measure: Mean (Standard Deviation); unit: EEG spike counts per minute
Groups:
- Dextromethorphan (DM)1 EEG Spike Counts at Baseline: Dextromethorphan(DM)I group received Dextromethorphan 0.25 mg/kg per day. The drug is given in two divided doses 12 hours apart for 6 months. EEG spike count for DM1 group measured at baseline.
- DM2 EEG Spike Counts at Baseline: DM2 group participants received Dextromethorphan 2.5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months. DM2 EEG spike counts at baseline.
- DM3 EEG Spike Counts at Baseline: DM3 group received Dextromethorphan 5mg/kg/day.
  The drug is given in two divided doses 12 hours apart for 6 months. EEG spike counts at baseline.
- DM1 EEG Spike Count at 6 Months: DM1 group received Dextromethorphan 0.25 mg/kg per day. The drug is given in two divided doses 12 hours apart for 6 months. EEG spike count for DM1 group measured at 6 months.
- DM2 EEG Spike Counts at 6 Months: DM2 group participants received Dextromethorphan 2.5 mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months. DM2 EEG spike counts at 6 months.
- DM3 EEG Spike Counts at 6 Months: DM3 group received Dextromethorphan 5mg/kg/day. The drug is given in two divided doses 12 hours apart for 6 months. EEG spike counts at 6 months.
Arm/Group | Dextromethorphan (DM)1 EEG Spike Counts at Baseline | DM2 EEG Spike Counts at Baseline | DM3 EEG Spike Counts at Baseline | DM1 EEG Spike Count at 6 Months | DM2 EEG Spike Counts at 6 Months | DM3 EEG Spike Counts at 6 Months
Number analyzed (Participants) | 13 | 12 | 8 | 13 | 12 | 8
EEG spike counts per minute | 44.22 (23.77) | 25.44 (18.6) | 40.67 (27.83) | 38.29 (30.24) | 27.58 (19.52) | 36.01 (23.29)
Statistical Analysis 1: Comparison: Dextromethorphan (DM)1 EEG Spike Counts at Baseline vs DM1 EEG Spike Count at 6 Months; Test type: Superiority or Other; p < 0.40, t-test, 2 sided
Statistical Analysis 2: Comparison: DM2 EEG Spike Counts at Baseline vs DM2 EEG Spike Counts at 6 Months; Test type: Superiority or Other; p < 0.62, t-test, 2 sided
Statistical Analysis 3: Comparison: DM3 EEG Spike Counts at Baseline vs DM3 EEG Spike Counts at 6 Months; Test type: Superiority or Other; p < 0.38, t-test, 2 sided

2. Secondary Outcome: Improvement in Receptive Language as Measured by the Mullen Scale.
Description: The Mullen Receptive language scale pre and 6 months post DM, measured as a change in the mean score of language, by age in months.
Time Frame: Change in mean between Initial and 6-month follow-up
Population: 25/35 enrolled participants completed the receptive language scale of the Mullen and underwent the analysis.
Measure: Mean (Standard Deviation); unit: age in months
Arm/Group | DM1( 0.25 mg/kg /Day) | DM2 (2.5 mg/kg/Day) | DM3 (5mg/kg/Day)
Number analyzed (Participants) | 10 | 8 | 7
age in months | 0 (2.94) | -0.44 (2.96) | 03 (2.45)

3. Secondary Outcome: Difference in SSI Mean Score at Six Months Compared to Baseline for Each Treatment Arm.
Description: The Screen for Social Interaction (SSI) is a 54-item parent/caregiver-report screening instrument that emphasizes reciprocal social interaction including joint attention skills. The items are positive (prosocial) and are scored on a four-point frequency scale (child displays the behavior "almost never" = 0 to "almost all the time" = 3). Thus lower scores reflect a slower or delayed development, and higher scores reflect more normative development. SSI total scores range from 0-162. There are no subscales. Difference in Screen for Social Interaction (SSI) mean scores between baseline and 6 months post-treatment for each treatment arm are reported.
Time Frame: Initial and 6 month followup
Population: Those who provided complete information only were included. Others did not provide adequate or complete information for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- DM1( 0.25 mg/kg /Day) SSI Baseline: Screen for Social Interaction (SSI) mean score at baseline for Dextromethorphan 0.25 mg/kg per day treatment arm.
- DM2 (2.5 mg/kg/Day)SSI Baseline: Screen for Social Interaction (SSI) mean score at baseline for Dextromethorphan 2.5 mg/kg/day treatment arm.
- DM3 (5mg/kg/Day) SSI Baseline: Screen for Social Interaction (SSI) mean score at baseline for Dextromethorphan 5mg/kg/day treatment arm.
- DM1( 0.25 mg/kg /Day) SSI 6 Months: DM1( 0.25 mg/kg /day)treatment arm Screen for Social Interaction (SSI) mean score at 6 months post-treatment.
- DM2 (2.5 mg/kg/Day) SSI 6 Months: DM2( 2.5 mg/kg /day)treatment arm Screen for Social Interaction (SSI) mean score at 6 months post-treatment.
- DM3 (5.0 mg/kg/Day) SSI 6 Months: DM3(5.0) mg/kg /day)treatment arm Screen for Social Interaction (SSI) mean score at 6 months post-treatment.
Arm/Group | DM1( 0.25 mg/kg /Day) SSI Baseline | DM2 (2.5 mg/kg/Day)SSI Baseline | DM3 (5mg/kg/Day) SSI Baseline | DM1( 0.25 mg/kg /Day) SSI 6 Months | DM2 (2.5 mg/kg/Day) SSI 6 Months | DM3 (5.0 mg/kg/Day) SSI 6 Months
Number analyzed (Participants) | 8 | 4 | 7 | 8 | 4 | 7
scores on a scale | 40.25 (18.59) | 70.00 (19.10) | 84.29 (17.51) | 48.63 (18.58) | 74.50 (22.78) | 88.29 (18.88)
Statistical Analysis 1: Comparison: DM1( 0.25 mg/kg /Day) SSI Baseline vs DM1( 0.25 mg/kg /Day) SSI 6 Months; Null hypothesis is that there would be no significant difference in social abilities as measured by the SSI score in this treatment group baseline to 6 months post-treatment; Test type: Superiority or Other; p < 0.10, ANOVA; Mean Difference (Final Values) = 8.38
Statistical Analysis 2: Comparison: DM2 (2.5 mg/kg/Day)SSI Baseline vs DM2 (2.5 mg/kg/Day) SSI 6 Months; Test type: Superiority or Other; p < 0.50, ANOVA; Mean Difference (Final Values) = 4.5
Statistical Analysis 3: Comparison: DM3 (5mg/kg/Day) SSI Baseline vs DM3 (5.0 mg/kg/Day) SSI 6 Months; Test type: Superiority or Other; p < 0.48, ANOVA; Mean Difference (Final Values) = 4.0

4. Secondary Outcome: Mean SSI Score for Total Subjects at Baseline and 6 Months
Description: Analysis of Difference in Mean Screen for Social Interaction (SSI) Score between 0-6 months for total sample (n=19).
Time Frame: 0-6 months
Population: 19 subjects (total sample) for whom complete data was available
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Total Sample SSI Mean Score at Baseline: Study Sample Screen for Social Interaction (SSI) mean core at baseline.
- Total Sample SSI Mean Score at 6 Months: Study Sample Screen for Social Interaction (SSI) mean score at 6 months post-treatment.
Arm/Group | Total Sample SSI Mean Score at Baseline | Total Sample SSI Mean Score at 6 Months
Number analyzed (Participants) | 19 | 19
scores on a scale | 62.737 (26.729) | 68.684 (25.987)
Statistical Analysis 1: Comparison: Total Sample SSI Mean Score at Baseline vs Total Sample SSI Mean Score at 6 Months; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 5.947

ADVERSE EVENTS:
Arm/Group | DM1( 0.25 mg/kg /Day) | DM2 (2.5 mg/kg/Day) | DM3 (5mg/kg/Day)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
The trial was terminated due to the FDA requiring a placebo controlled trial instead of the ongoing open label trial. As recruitment was delayed,the total number of participants was also less than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No